CLINICAL TRIAL: NCT06234436
Title: Plasma Dilution and Infusion to Improve Cognition in Mild Cognitive Impairment (MCI)
Acronym: ADDITION-MCI
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Oslo University Hospital (Other)
Collaborators: Impetus Grants (EIN: 87-1540960) (Unknown); The National Association for Public Health, Norway (Other Government); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Arne Vasli Lund Søraas, PI, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 520697
Record Dates: First submitted 2023-12-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a safety and feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasma exchange (Experimental): 1-20 plasma exchanges.
  Interventions: Biological: Plasma exchenge

INTERVENTIONS:
Biological: Plasma exchenge — Plasma exchange will be conducted. The substitution fluid will be plasma from ha healthy donor.

SUMMARY:
In the ADDITION-MCI project, patients with a diagnosis of mild cognitive impairment probably caused by Alzheimer's disease will receive plasma exchange.

DETAILED DESCRIPTION:
Repeated plasma exchanges will be conducted, and cognitive outcomes will be measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Alzheimer's Disease

MoCA score < 27 and >17

Able to give informed consent as judged by the doctor setting the AD diagnosis and study doctor.

At least one biomarker of the AT(N)-classification system supporting the diagnosis

Expected to live more than five years at inclusion by the study doctor.

Exclusion Criteria:

Known IgA deficiency

Known severe protein S depletion

Previous severe allergic reaction after transfusion of a blood product

Known heart failure

Known liver failure

Known kidney failure

Previous cancer <10 years.

Not deemed able to participate by the study staff

Other severe chronic diseases, interfering with the TPE-procedure

Ongoing infections

Other unresolved medical conditions

Known coagulopathies

Fulfilling ICD-10 criteria for dementia at baseline, as evaluated by the evaluating physician.

Peripheral veins not expected to be suitable for repeated venous access procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Up to 4 years
  Safety of the intervention in the patient group measured as number and severity of adverse events.
  This will be evaluated as the number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) Test for Dementia | 2 months
  Change from baseline to after completion of all procedure cycles
Change in Montreal Cognitive Assessment (MoCA) Test for Dementia | 6 months
  Change from baseline to after the procedure
Change in Montreal Cognitive Assessment (MoCA) Test for Dementia | 12 months
  Change from baseline to after the procedure
Change in Montreal Cognitive Assessment (MoCA) Test for Dementia | 24 months
  Change from baseline to after the procedure
Change in Montreal Cognitive Assessment (MoCA) Test for Dementia | 48 months
  Change from baseline to after the procedure
Burden of participation questionnaire sum score | 2 months
  At the end of the procedure
Change in IL10 from baseline | 2 months
  Change in IL10
Change in IL10 from baseline | 6 months
  Change in IL10
Change in IL6 from baseline | 2 months
  Change in IL6
Change in IL6 from baseline | 6 months
  Change in IL6
Change in grip strength from baseline | 2 months
  Change in grip strength from baseline
Change in grip strength from baseline | 6 months
  Change in grip strength from baseline
Change in grip strength from baseline | 12 months
  Change in grip strength from baseline
Change in grip strength from baseline | 24 months
  Change in grip strength from baseline
Change in grip strength from baseline | 48 months
  Change in grip strength from baseline
Change in the CERAD 10-word test performance from baseline | 2 months
  Change in the CERAD 10-word test performance from baseline
Change in the CERAD 10-word test performance from baseline | 6 months
  Change in the CERAD 10-word test performance from baseline
Change in the CERAD 10-word test performance from baseline | 12 months
  Change in the CERAD 10-word test performance from baseline
Change in the CERAD 10-word test performance from baseline | 24 months
  Change in the CERAD 10-word test performance from baseline
Change in the CERAD 10-word test performance from baseline | 48 months
  Change in the CERAD 10-word test performance from baseline
Change in the trail making test A or B (as appropriate) time from baseline | 2 months
  Change in the trail making test A or B (as appropriate) time from baseline
Change in the trail making test A or B (as appropriate) time from baseline | 6 months
  Change in the trail making test A or B (as appropriate) time from baseline
Change in the trail making test A or B (as appropriate) time from baseline | 12 months
  Change in the trail making test A or B (as appropriate) time from baseline
Change in the trail making test A or B (as appropriate) time from baseline | 24 months
  Change in the trail making test A or B (as appropriate) time from baseline
Change in the trail making test A or B (as appropriate) time from baseline | 48 months
  Change in the trail making test A or B (as appropriate) time from baseline
Change in IQCODE from baseline | 2 months
  Measured at the nearest next-of-kin
Change in IQCODE from baseline | 6 months
  Measured at the nearest next-of-kin
Change in IQCODE from baseline | 12 months
  Measured at the nearest next-of-kin
Change in IQCODE from baseline | 24 months
  Measured at the nearest next-of-kin
Change in IQCODE from baseline | 48 months
  Measured at the nearest next-of-kin
Change in 4 meter walk test from baseline | 2 months
Change in 4 meter walk test from baseline | 6 months
Change in 4 meter walk test from baseline | 12 months
Change in 4 meter walk test from baseline | 24 months
Change in 4 meter walk test from baseline | 48 months

OTHER OUTCOMES:
Change in DNA methylation age GrimAge2 from baseline | 6 months
  Epigenetic measurement
Proteomic profile | 12 months
  Comparison of the proteomic profile at baseline and the proteomic profile at 12 months. The profile will be measured using SomaLogic assays and in this endpoint the concentration of each protein at baseline will be compared to the concentration at 12 months.
Single cell RNA seq | 6 months
Change in EQ5D | 12 months
  The EQ5D questionnaire will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
We will attempt to share IDP within the European GDPR rules.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Before data analysis and publication
Access Criteria: On request to the study contact.